CLINICAL TRIAL: NCT01495806
Title: Glucomannn for the Treatment of Abdominal Pain-related Functional Gastrointestinal Disorders in Childhood Randomized Double Blind Placebo Controlled Trial
Brief Title: Glucomannan for the Treatment of Abdominal Pain-related Functional Gastrointestinal Disorders in Childhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrea Horvath-Stolarczyk, dr, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010
Record Dates: First submitted 2011-07-12; First posted 2011-12-20 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: functional dyspepsia; irritable bowel syndrome; functional abdominal pain
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucomannan (Experimental): 5 g 2x 10 day
  Interventions: Drug: Glucomannan
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Glucomannan — 2 x 5g
  Arms: Glucomannan
Drug: placebo — glucose 5 g
  Arms: Placebo

SUMMARY:
Background: Functional abdominal pain disorders (FAPD) are common in school-aged children; however, there is no reliable treatment.

Aim: To determine the efficacy and safety of glucomannan for treating FAPD in children.

Trial Setting: Department of Pediatrics, The Medical University of Warsaw.

Intervention: Patients will be enrolled in a double-blind, randomized controlled trial in which they will receive either glucomannan (10g) or placebo for 4 weeks.

DETAILED DESCRIPTION:
According to the Rome III criteria, abdominal pain-related functional gastrointestinal disorders (FGD) in children may be categorised as functional dyspepsia (FD), irritable bowel syndrome (IBS), abdominal migraine and functional abdominal pain (FAP). Because of their obscure pathophysiology, management of abdominal pain-related FGD remains difficult, prompting interest in new and safe treatment options.Glucomannan is a prebiotic which is nondigestible food ingredients that beneficially affect the host by selectively stimulating the growth and ⁄ or activity of bacteria already resident in the colon. Up to now there has been published one randomized controlled trial which showed that treatment with the prebiotic (trans-galactooligosaccharide), which induced qualitative changes in the faecal flora, was associated with significant changes in stool consistency, flatulence, composite scores (abdominal pain ⁄ discomfort, bloating ⁄ distension and bowel movement difficulty) as well as subjective global assessment values in adult patients with irritable bowel syndrome. These findings suggest that the prebiotics has a potential as a therapeutic agent in functional gastrointestinal disorders.

Methods Patients will be recruited from children referred to the Department of Pediatrics, The Medical University of Warsaw. Each potentially eligible patient will be evaluated by a full review of their clinical history and physical examination. Subjects will receive a questionnaire to record the frequency and severity of pain, drug use and any symptoms they considered important for the last 4 weeks. Patients will be considered for study inclusion, if they will be 8-18 years of age and will have an abdominal pain - related disorder (i.e. (functional dyspepsia, irritable bowel syndrome or functional abdominal pain ( FD or IBS or FAP) classified according to the Rome III diagnostic criteria. Patients with organic gastrointestinal disease (as established by medical history, complete blood count, urinalysis, stool examination for occult blood, ova and parasites, blood chemistries, abdominal ultrasound, breath hydrogen testing and endoscopy, if needed),other chronic disease, growth failure will be excluded from the study. A total of 90 children who will fulfill the Rome III criteria for functional dyspepsia (FD), or irritable bowel syndrome (IBS), or functional abdominal pain (FAP) will be enrolled in a double-blind, randomized controlled trial in which they will received either glucomannan 10g (n = 45), or placebo (n = 45) for 4 weeks. At the end of the study patients will fulfill the questionnaire assessing the outcome measures. The primary outcome measure is treatment success defined as no pain (a relaxed face, score of 0, on the Faces Pain Scale) at the end of the intervention. The secondary outcome measures are (i) improvements in self-reported severity of pain defined as a change in by at least two faces scores measured on the Faces Pain Scale; (ii) self-reported frequency of pain during the preceding month; (iii) use of medication for abdominal pain and (iv) school absenteeism because of abdominal pain.(v)adverse events during the study period.

Statistical Methods The statistical analyses will be conducted with StatsDirect. The Mann-Whitney U test will be used to compare the means of continuous variables if non-normal distribution will be assessed. Proportions will be compared with the Fisher exact test. The difference in study groups was considered significant when the P value will be <.05. the results of this study will be analyzed on the basis of intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* abdominal pain related disorder (functional dyspepsia, irritable bowel syndrome or functional abdominal pain (FAPS) diagnosed according to Rome III criteria.

Exclusion Criteria:

* organic gastrointestinal disease (as established by medical history, complete blood count, urinalysis, stool examination for occult blood, ova and parasites, blood chemistries, abdominal ultrasound, breath hydrogen testing and endoscopy, if needed)
* other chronic disease
* growth failure

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
number of patients with no abdominal pain at the end of the study | 4 weeks (study period)

SECONDARY OUTCOMES:
number of patients with improvement in self-reported severity of pain | 4 weeks study period
  improvement in self-reported severity of pain is defined as at least two Faces Pain Score improvement at the end of the study compared to the baseline
number of patients suffered from abdominal pain < 1/week | 4 weeks (during the study period)
  self reported with questionnaire
number of patients who used medication for abdominal pain | 4 weeks study period
  self reported assessed with questionnaire
number of patients who lost min.1 school day because of abdominal pain | 4 weeks (study period)
  self reported with the questionnaire
Number of participants with adverse events as a measure of safety and tolerability | participants will be followed for the duration of h an expected average of 4 weeks - study period
  self assessed with the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Horvath, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Dpt of Pediatrics Warsaw Medical University, Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Horvath A, Dziechciarz P, Szajewska H. Glucomannan for abdominal pain-related functional gastrointestinal disorders in children: a randomized trial. World J Gastroenterol. 2013 May 28;19(20):3062-8. doi: 10.3748/wjg.v19.i20.3062. PMID 23716985